CLINICAL TRIAL: NCT06938178
Title: High-Density EEG-MEG-wearable EEG: Comparison of Quantitative Electroencephalographic Indicators as Neurophysiological Markers of Effectiveness of Mindfulness Therapy in Addition to Standard Treatment in Patients With High-frequency Episodic Migraine
Acronym: MindMEEG
Status: Recruiting | Type: Observational
Sponsor: Fondazione I.R.C.C.S. Istituto Neurologico Carlo Besta (Other)
Responsible Party: Sponsor
Other Study IDs: MindMEEG
Record Dates: First submitted 2025-04-04; First posted 2025-04-22 (Actual); Last update posted 2025-04-22 (Actual); Status verified 2025-04

CONDITIONS: Migraine; Migraine Disease; High Frequency Episodic Migraine
Keywords: Migraine; MEG; Mindfulness; Wearable EEG
MeSH Terms: conditions — Migraine Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Group Mindfulness treatment: group undergoing 8 weeks of Mindfulness treatment and unchanged drug therapy
  Interventions: Other: Mindfulness treatment
- Group Standard of care: group re-evaluated after 8 weeks without any additional intervention and with unchanged drug therapy.

INTERVENTIONS:
Other: Mindfulness treatment — The Mindfulness treatment will consist of a series of 8 weekly meetings in small groups . An experienced therapist will guide patients and during the sessions they will be encouraged to close their eyes, assume a relaxed posture, focus on breathing and the present moment in order to improve awareness of mental and bodily sensations. Patients will also be encouraged to add a regular, practice at home of about 10 minutes to the group treatment. If necessary, patients in both groups can take the medication they normally take for acute events. These occurrences will be reported in the headache diary given to each subject. Before conducting the study protocol, the investigator will explain the study to each participant and collect a signed copy of the written informed consent. All participants will undergo a clinical, neurophysiological and neuropsychological evaluation before the first session and after the last. In both groups, the usual drug therapies in case of crisis will be allowed.
  Groups: Group Mindfulness treatment

SUMMARY:
Recent studies suggest that Mindfulness may be an effective treatment for migraine, reducing the frequency of attacks, depression, anxiety and improving quality of life. However, the pathophysiological mechanisms underlying the effectiveness are not yet fully known. The identification of neurophysiological markers may help to better understand the mechanisms on which Mindfulness acts in migraine sufferers and to develop increasingly targeted and personalized Mindfulness interventions to optimize migraine treatment. The main objective of the study is to identify neurophysiological indicators of effectiveness of Mindfulness treatment in patients with migraine without high-frequency aura with clinically available devices (MEG and hdEEG). Another goal is to recognize the indicators also in the signal acquired with wearable devices in home use (wEEG). Finally, another goal will be to study the relationship between the identified neurophysiological markers and the change in neuropsychological test scores.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients will be included who fulfil the ICHD-3 criteria [8] for HFEM, code 1.3-Chronic Migraine (characteristics similar to CM but with a frequency of 8-14 migraine days per month) with stable therapy in the 3 months prior to the start of Mindfulness treatment. If the therapy is changed during the screening visit, the patient will wait 3 months before starting Mindfulness treatment.

Exclusion Criteria:

* in the presence of psychiatric comorbidities in the psychotic area, reported in the history or assessed by the clinician
* if pregnant
* in the presence of secondary headache comorbidities (e.g. idiopathic intracranial hypertension)
* if they have undergone symptomatic abuse detoxification at least twice in the previous two years
* if they have already undergone any kind of treatment with Mindfulness or meditation techniques

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Adult patients will be included who fulfil the ICHD-3 criteria for high-frequency migraine (8-14 migraine days per month) with stable therapy in the 3 months prior to study participation. If the therapy is changed during the screening visit, the patient will wait 3 months before being included in the study. Patients will be excluded in in the presence of psychiatric comorbidities in the psychotic area, reported in the history or assessed by the clinician, if pregnant, in the presence of secondary headache comorbidities (e.g. idiopathic intracranial hypertension), if they have undergone symptomatic abuse detoxification at least twice in the previous two years and if they have already undergone any kind of treatment with Mindfulness or meditation techniques
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2024-04-23 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Correlation between neurophysiological indicators and clinical outcome | through study completion, an average of 2 years
  The primary endpoint is the correlation between change in quantitative neurophysiological indices from MEG and hdEEG and change in attack characteristics (monthly frequency, intensity, duration, and use of symptomatic medication) of migraine without aura after treatment with Mindfulness. Quantitative indices of brain activity will include frequency and amplitude of the peaks in the canonical bands (delta: 1-4 Hz, theta: 4-8 Hz, alpha: 8-12 Hz, beta: 13-30 Hz), relative power in the canonical bands, power ratio (DAR: delta/alpha power ratio; DTABR: (delta + theta)/(alpha + beta) power ratio, BSI: brain symmetric index).

SECONDARY OUTCOMES:
Correlation between neurophysiological indicators calculated with different types of device | through study completion, an average of 2 years
  A secondary outcome is the correlation between the quantitative neurophysiological indices (frequency and amplitude of peaks and relative power in canonical bands, DAR, DTABR, BSI) obtained from signals acquired with clinical high-density instrumentation (hdEEG and MEG) and the same indices obtained from signals acquired with low-density instrumentation (wEEG)
Correlation between neurophysiological indicators and neuropsychological scores | through study completion, an average of 2 years
  A secondary outcome is the correlation between variation in quantitative neurophysiological indices (frequency and amplitude of peaks and relative power in canonical bands, DAR, DTABR, BSI) assessed with both high-density and low-density instrumentations and variation in neuropsychological test scores (Migraine-Specific Quality of Life Questionnaire 2.1, Pain Catastrophizing Scale, General Self Efficacy Scale, Mindful Attention Awareness Scale, Multidimensional Assessment of Interoceptive Awareness, Beck Depression Inventory II, State-Trait Anxiety Inventory-Y)

CONTACTS AND LOCATIONS:
Overall Officials: Paola Lanteri, MD, Principal Investigator — Fondazione IRCCS Istituto Neurologico Carlo Besta
Locations (1):
- Fondazione IRCCS Istituto Neurologico C. Besta, Milan, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tang YY, Tang R, Rothbart MK, Posner MI. Frontal theta activity and white matter plasticity following mindfulness meditation. Curr Opin Psychol. 2019 Aug;28:294-297. doi: 10.1016/j.copsyc.2019.04.004. Epub 2019 Apr 18. PMID 31082635
- [Background] Grazzi L, D'Amico D, Guastafierro E, Demichelis G, Erbetta A, Fedeli D, Nigri A, Ciusani E, Barbara C, Raggi A. Efficacy of mindfulness added to treatment as usual in patients with chronic migraine and medication overuse headache: a phase-III single-blind randomized-controlled trial (the MIND-CM study). J Headache Pain. 2023 Jul 14;24(1):86. doi: 10.1186/s10194-023-01630-0. PMID 37452281
- [Background] Grazzi L, Montisano DA, Raggi A, Rizzoli P. Feasibility and effect of mindfulness approach by web for chronic migraine and high-frequency episodic migraine without aura at in adolescents during and after COVID emergency: preliminary findings. Neurol Sci. 2022 Sep;43(9):5741-5744. doi: 10.1007/s10072-022-06225-2. Epub 2022 Jul 4. PMID 35788839
- [Background] Sansone E, Grazzi L, Raggi A, Leonardi M, D'Amico D. Mindfulness as an add-on treatment for patients with chronic migraine and medication overuse: a preliminary analysis. Neurol Sci. 2020 Dec;41(Suppl 2):469-471. doi: 10.1007/s10072-020-04662-5. No abstract available. PMID 32845485
- [Background] Seng EK, Singer AB, Metts C, Grinberg AS, Patel ZS, Marzouk M, Rosenberg L, Day M, Minen MT, Lipton RB, Buse DC. Does Mindfulness-Based Cognitive Therapy for Migraine Reduce Migraine-Related Disability in People with Episodic and Chronic Migraine? A Phase 2b Pilot Randomized Clinical Trial. Headache. 2019 Oct;59(9):1448-1467. doi: 10.1111/head.13657. Epub 2019 Sep 26. PMID 31557329
- [Background] Harris P, Loveman E, Clegg A, Easton S, Berry N. Systematic review of cognitive behavioural therapy for the management of headaches and migraines in adults. Br J Pain. 2015 Nov;9(4):213-24. doi: 10.1177/2049463715578291. PMID 26526604
- [Background] Ailani J, Burch RC, Robbins MS; Board of Directors of the American Headache Society. The American Headache Society Consensus Statement: Update on integrating new migraine treatments into clinical practice. Headache. 2021 Jul;61(7):1021-1039. doi: 10.1111/head.14153. Epub 2021 Jun 23. PMID 34160823